CLINICAL TRIAL: NCT00960791
Title: An Open, Single-centre, Single Group, Phase I Study to Assess the Absorption, Distribution, Metabolism and Excretion (ADME) of AZD1656 After Oral Administration of 14C-labelled AZD1656 to Type II Diabetes Mellitus Patients
Brief Title: Study to Assess the Absorption, Distribution, Metabolism and Excretion of AZD1656 in Type 2 Diabetes Mellitus (T2DM)
Acronym: ADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00008
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II diabetes mellitus; absorption; distribution; metabolism; excretion; 14C-labelled
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- 1 (Experimental): 14C-labelled AZD1656
  Interventions: Device: AZD1656

INTERVENTIONS:
Device: AZD1656 — Oral single dose

SUMMARY:
The purpose of the study is to evaluate the absorption, distribution, metabolism and excretion of AZD1656 after administration of a single oral dose of 14C-labelled AZD1656 solution in male Type 2 Diabetes Mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Male type II diabetes patients diagnosed for more than 5 years and aged between 35 and 65 years.
* Subjects treated with metformin alone or metformin and one other oral anti-diabetic drug.
* Subjects should have FPG in the range of 6.0 to 11.0 mmol/L at screening and HbA1c less than 10% (HbA1c value according to international DCCT standard).

Exclusion Criteria:

* History of ischemic heart disease, stroke, transient ischemic attack or symptomatic peripheral vascular disease.
* Renal dysfunction.
* Use of insulin, glitazones, warfarin and amiodarone within 3 months before enrolment and use of potent CYP450 inhibitors, e.g., ketoconazole and macrolide antibiotics within 14 days before administration of IP.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-07; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Total recovery of radioactive dose, rate and routes of excretion of total radioactivity, metabolic pattern and metabolic profile, and PK variables of AZD1656 (AUC, Cmax, tmax, t1/2, Total Ae, CL/F and CLR) | One blood sample for analysis of plasma concentrations of AZD1656 taken on several days during the treatment period. A full PK profile for AZD1656 will also be taken on the last day of treatment

SECONDARY OUTCOMES:
Safety variables: Adverse Events (AEs), Blood pressure (BP), pulse, ECG and safety laboratory variables, glucose quick test | Frequent measurements during the study period
Plasma Glucose | Plasma Glucose will be measured twice daily during residential period

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof.,, Study Director — AstraZeneca R&D Mölndal, SE-431 83 Mölndal, Sweden; Emeline Ramos, MD, Principal Investigator — Clinical Pharmacology Unit (CPU)AstraZeneca R&D Alderley ParkMacclesfield, Cheshire SK10 4TG, UK
Locations (2):
- United States (2):
  - Research Site, San Diego, California
  - Research Site, San Antonio, Texas